CLINICAL TRIAL: NCT06790420
Title: RITUXIMAB BS Intravenous Infusion 100mg・500mg [Pfizer] Post-marketing Database Study
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3281009
Record Dates: First submitted 2025-01-09; First posted 2025-01-24 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma
Keywords: Lymphoma; Rituximab; Infection
MeSH Terms: conditions — Lymphoma; Infections | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: patients treated with Rituximab Pfizer
  Interventions: Drug: Rituximab Pfizer
- Comparative group: patients treated with Rituxan
  Interventions: Drug: Rituxan

INTERVENTIONS:
Drug: Rituximab Pfizer — For the acute therapy, Rituximab is administrated once a week up to 8 times and for maintenance therapy, it is administrated every 8 weeks up to 12 times
  Groups: Exposed group
Drug: Rituxan — For the acute therapy, Rituximab is administrated once a week up to 8 times and for maintenance therapy, it is administrated every 8 weeks up to 12 times
  Groups: Comparative group

SUMMARY:
To evaluate the incidence of the outcomes for the safety specifications in patients of Medical Data Vision database in Japan diagnosed with CD20 positive B-cell non- Hodgkin's lymphoma who were treated with Rituximab Pfizer to compare it with outcomes in patients who were treated with Rituxan from 01 January 2020 through 31 December 2024

ELIGIBILITY:
Inclusion Criteria:

1. Have prescription of Rituximab Pfizer or Rituxan within the enrollment period (Index Date: first prescription date within the enrollment period).
2. Have diagnosis of CD20 positive B-cell non- Hodgkin's lymphoma on the index month or within 6 months before index date
3. Have at least 6 months of Look back period and at least one medical record prior to 7 months before the Index date.
4. Have not prescription of Rituximab product before index date(Comparative Analysis Set only).

Exclusion Criteria:

1. Have any diagnosis of other indications of rituximab products other than CD20 positive B-cell non- Hodgkin's lymphoma before index date .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals who have a diagnosis of CD20 positive B-cell non- Hodgkin's lymphoma and treated with Rituximab Pfizer and Rituxan
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Incidence of infections which requires procedures, medication or hospitalization | From index date up to 180 days after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of continuous treatment plus 180 days risk window, death, loss to follow up or the end of study period

SECONDARY OUTCOMES:
Incidence of 'pancytopenia, leukocytopenia, Neutropenia, agranulocytosis, thrombocytopenia' | From index date up to 180 days after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of continuous treatment plus 180 days risk window, death, loss to follow up or the end of study period
Incidence of Infusion reactions | From index date up to next day after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of risk window which is until next day after last dose, death, or the end of study period.
Incidence of hepatic function disorder, jaundice | From index date up to 180 days after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of continuous treatment plus 180 days risk window, death, loss to follow up or the end of study period
Incidence of cardiac disorder | From index date up to 180 days after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of continuous treatment plus 180 days risk window, death, loss to follow up or the end of study period
Incidence of gastrointestinal perforation/obstruction | From index date up to 180 days after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of continuous treatment plus 180 days risk window, death, loss to follow up or the end of study period
Incidence of hypotension | From index date up to next day after last dose
  until the first incidence of an event, date of switch to another Rituximab product, the end of risk window which is until next day after last dose, death, or the end of study period.
Incidence of development of malignant tumor | From index date up to maximum of 5 years (the end of the study period)
  follow until the first incident event, death, end of the study period, or loss to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.